CLINICAL TRIAL: NCT02329145
Title: Renal Denervation in Patients With Chronic Heart Failure and Resynchronization Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Aleksander Kusiak, MD, PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204069
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Heart Failure
Keywords: renal denervation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (Experimental): Renal denervation
  Interventions: Procedure: renal denervation
- Observational (No Intervention)

INTERVENTIONS:
Procedure: renal denervation
  Arms: Active treatment

SUMMARY:
Chronic heart failure is becoming more and more common disease and activation of sympathetic nervous system plays a crucial role in its development. There is some data allowing to suspect that one of the new treatment methods- renal denervation, also in patients with chronic heart failure may lead to decrease of systemic activity sympathetic nervous system and, as a consequence, to decrease of disease progression. The research hypothesis is whether renal denervation in case of symptomatic heart failure, even the optimal treatment therapy is used (including resynchronization therapy), is contributing to the improvement in parameters of neurohormonal activation, hemodynamics and clinical patient status. The aim of the study is to obtain a new knowledge concerning renal denervation in chronic heart failure, So far only very limited data- mostly case reports- are available in this study area.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 year
2. heart failure patients NYHA Class II - IV
3. implanted resynchronization pacemaker according to current european guidelines at least 6 months earlier
4. symptoms of heart failure even on optimal pharmacological therapy including resynchronization therapy (lack of improvement within dyspnoea and exercise tolerance after the procedure)
5. left ventricular ejection function ≤ 35%
6. glomerular filtration rate (eGFR according to MDRD formula ≥ 30 mL/min/1.73m2)
7. patient informed consent for participation in the study

Exclusion Criteria:

1. renal artery anatomy not eligible for denervation (at least 4 mm diameter, 20 mm in length)
2. history of prior renal artery intervention
3. single functioning kidney
4. clinic systolic BP < 110mmHg
5. pregnancy
6. acute coronary syndrome or cerebrovascular event within last 3 months
7. serious medical conditions which may adversely affect safety- clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders (thrombocytopenia, hemophilia, or significant anemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalizations due to heart failure worsening. | one year
Change in NYHA class. | one year
Change in 6 minute walk test distance. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Ist Department of Cardiology, Interventional Electrocardiology and Hypertension, Krakow, Malopolska, Poland